CLINICAL TRIAL: NCT03205514
Title: Multimodality Investigation of Intermediate Culprit Lesion With Negative Fractional Flow Reserve in Patients With no ST-segment Elevation Acute Coronary Syndrome.
Brief Title: Multimodality Investigation of Intermediate Culprit Lesion With Negative FFR in NSTE-ACS
Acronym: SHERLOCK
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, University Hospital of Ferrara
Other Study IDs: 160487
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSTE-ACS with intermediate stenosis and negative FFR: Patients hospitalized because of an acute coronary syndrome without ST segment elevation and with intermediate culprit lesion with negative fractional flow reserve evaluation (>0.80).
  Interventions: Diagnostic Test: NSTE-ACS with intermediate stenosis and negative FFR

INTERVENTIONS:
Diagnostic Test: NSTE-ACS with intermediate stenosis and negative FFR — Patients will undergo intracoronary imaging evaluation with IVUS-NIRS and OCT, endothelial function and inflammatory state evaluation.

SUMMARY:
Ten-fifteen percent of acute coronary syndromes without ST-segment elevation (NSTE-ACS) are caused by intermediate lesions without signs of unstable plaque. In this subset of patients, fractional flow reserve (FFR) has some drawbacks and may not be always able to predict outcome, especially when negative (above 0.80). In this particular nique of patients, advanced imaging techniques are suggested by International guidelines. However, it is actually unknown how these techniques may impact treatment strategies. With the present study, the investigators want to characterize the mechanism of disease in this particular subset of patients through multimodality imaging (intravascular ultrasound-near infrared spectroscopy (IVUS-NIRS), optical coherence tomography (OCT)) in order to understand the proper treatment.

DETAILED DESCRIPTION:
Acute coronary syndrome without ST-segment elevation (NSTE-ACS) is by far the most frequent acute coronary syndrome (ACS) in the western world. In most of the cases, it is caused by a clearly identifiable culprit lesion, configuring a significant angiographic stenosis (>70%), with flux limitation and typical aspects of unstable plaque (thrombosis). In these cases, the one and only treatment is stent implantation. In a small percentage of patients (10-15%), NSTE-ACS is caused by an angiographically intermediate lesion (40-70%). This lesion is identifiable as culprit, but without the typical signs of unstable plaque.

In patients with stable coronary artery disease (SCAD) presenting with this type of lesion, fractional flow reserve (FFR) is the actual gold-standard for ischemic burden evaluation. Several studies showed that if FFR value is ≤0.80, the treatment with percutaneous coronary intervention (PCI) is associated with a significant reduction of hard cardiovascular events. When FFR is negative (>0.80), optical medical therapy showed a better outcome when compared to percutaneous intervention. In NSTE-ACS, FFR evaluation of intermediate lesions is still mandatory, as a recent study showed a better outcome in patient with positive fractional flow reserve treated invasively with stenting compared to patients treated solely based on angiography (1). When FFR is negative, several authors and studies suggest that further imaging techniques are needed. In this subgroup of patients with intermediate stenosis without angiographic evidence of plaque rupture, European Guidelines (2) suggest utilization of intravascular ultrasound-near infrared spectroscopy (IVUS-NIRS) or optical coherence tomography (OCT) in order to better characterize the culprit plaque. At the same time, the therapeutic strategy is left to the operator's discretion: some implant a stent in order to reduce occurrence of future events, while some others leave the patient in optical medical therapy without stent implantation. Moreover, in these patients, it is still unclear the pathophysiology of the disease leading to ACS. In the last years, researchers focused their attention on plaque erosion, deemed to be responsible for most of these NSTE-ACS (3). An imaging study evaluated the incidence of plaque erosion in patients with ACS (4). This study enrolled an heterogeneous group of patients, evaluated with a single imaging technique (OCT).

Based on these background, the investigators hypothesized to perform a prospective single-center data registry on this highly selected subgroup of patients: NSTE-ACS with culprit intermediate lesion with negative FFR evaluation.

Investigators will enroll consecutive patients with NSTE-ACS with a culprit intermediate stenosis between 40 and 70% and in whom FFR evaluation will result negative (>0.80). In these patients, the operator will perform IVUS-NIRS and OCT and a blood sample to evaluate endothelial function as per our previous experience (5). The study has no control group. Endothelial function and inflammatory state will be evaluated in all patients and will be compared to those obtained by patients enrolled in the NATHAN NEVER study (NCT02519608, Study ID: 150497)(5).

Aim of the present study is to understand whether in this group of patient endothelial function is impaired and which information is given by intracoronary imaging (presence of plaque erosion). The present study is a prospective data collection. Thus, a formal sample size calculation is not applicable. Contemporaneously, for pilot studies, at least 30 patients are recommended (6).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of no-ST elevation-acute coronary syndrome
* clinical indication to coronary artery angiography
* angiographic documentation of intermediate lesion (40%-70%) with anterograde TIMI 3 flow eligible for FFR evaluation
* negative FFR evaluation (>0.80)

Exclusion Criteria:

* cardiogenic shock
* any indication to stent treatment for lesion
* previous stent implantation on the target vessel
* left main disease
* massive thrombus presence in the culprit vessel
* life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSTE-ACS patients with intermediate culprit lesion (40-70%) and negative FFR (>0.80).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Plaque erosion incidence | intra-procedure
  OCT-erosion: evidence of thrombotic material, irregular luminal surface without evidence of plaque fissure in multiple adjacent frames.
  IVUS/NIRS erosion: evidence of thrombotic material, irregular luminal surface without evidence of plaque fissure in multiple adjacent frames with lipid core burden index lower than the validated cutoff for unstable plaque (LCBI 4mm<400).

SECONDARY OUTCOMES:
Incidence of intermediate lesions with negative FFR in NSTE-ACS | intra-procedure
  Incidence of intermediate lesions with negative FFR in the whole population of NSTE-ACS
Vessel Lipid burden | intra-procedure
  Vessel Lipid burden at IVUS-NIRS evaluation (total LCBI) in patients with intermediate plaque and negative FFR
Plaque Lipid burden | intra-procedure
  Plaque Lipid burden at IVUS-NIRS evaluation (max LCBI 4 mm) in patients with intermediate plaque and negative FFR
Apoptosis rate in HUVEC | intra-procedure
  Rate of apoptosis in human umbilical vein endothelial cells (HUVEC) incubated with serum from patients enrolled in the study.
NO intracellular levels | intra-procedure
  Modulation of intracellular levels of nitric oxid (NO) in HUVECs treated with serum from patients enrolled in the study
ROS production | intra-procedure
  Intracellular levels of reactive oxygen species (ROS) in peripheral blood mononuclear cells (PBMCs) isolated from patients enrolled in the study
Inflammation markers levels | intra-procedure
  Values of the most important inflammation cytokines (hs-PCR, fibrinogen, IL-6, IL-1Ra, TNF-alpha)
Ischemic adverse events | 1 year
  Cumulative incidence of ischemic adverse events (death, myocardial infarction, stent thrombosis).

CONTACTS AND LOCATIONS:
Overall Officials: Simone Biscaglia, MD, Principal Investigator — Ferrara University Hospital
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Layland J, Oldroyd KG, Curzen N, Sood A, Balachandran K, Das R, Junejo S, Ahmed N, Lee MM, Shaukat A, O'Donnell A, Nam J, Briggs A, Henderson R, McConnachie A, Berry C; FAMOUS-NSTEMI investigators. Fractional flow reserve vs. angiography in guiding management to optimize outcomes in non-ST-segment elevation myocardial infarction: the British Heart Foundation FAMOUS-NSTEMI randomized trial. Eur Heart J. 2015 Jan 7;36(2):100-11. doi: 10.1093/eurheartj/ehu338. Epub 2014 Sep 1. PMID 25179764
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Libby P, Pasterkamp G. Requiem for the 'vulnerable plaque'. Eur Heart J. 2015 Nov 14;36(43):2984-7. doi: 10.1093/eurheartj/ehv349. Epub 2015 Jul 22. No abstract available. PMID 26206212
- [Background] Jia H, Abtahian F, Aguirre AD, Lee S, Chia S, Lowe H, Kato K, Yonetsu T, Vergallo R, Hu S, Tian J, Lee H, Park SJ, Jang YS, Raffel OC, Mizuno K, Uemura S, Itoh T, Kakuta T, Choi SY, Dauerman HL, Prasad A, Toma C, McNulty I, Zhang S, Yu B, Fuster V, Narula J, Virmani R, Jang IK. In vivo diagnosis of plaque erosion and calcified nodule in patients with acute coronary syndrome by intravascular optical coherence tomography. J Am Coll Cardiol. 2013 Nov 5;62(19):1748-58. doi: 10.1016/j.jacc.2013.05.071. Epub 2013 Jun 27. PMID 23810884
- [Background] Campo G, Vieceli Dalla Sega F, Pavasini R, Aquila G, Gallo F, Fortini F, Tonet E, Cimaglia P, Del Franco A, Pestelli G, Pecoraro A, Contoli M, Balla C, Biscaglia S, Rizzo P, Ferrari R. Biological effects of ticagrelor over clopidogrel in patients with stable coronary artery disease and chronic obstructive pulmonary disease. Thromb Haemost. 2017 Mar 23;117(6):1208-1216. doi: 10.1160/TH16-12-0973. Epub 2017 Mar 23. PMID 28331925
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396